CLINICAL TRIAL: NCT00955201
Title: Exercise-Facilitated NeuroRehabilitation in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: B6954-R; I01RX000130 (NIH)
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Neuropathy
Keywords: diabetes mellitus; diabetic neuropathies; Aerobic Exercise; Exercise Therapy; electromyography; United States Veterans
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (No Intervention): Sedentary Control Group
- Arm 2 (Experimental): Aerobic Exercise Group
  Interventions: Behavioral: Exercise
- Arm 3 (Experimental): Isokinetic Strength Exercise Group
  Interventions: Behavioral: Exercise
- Arm 4 (Experimental): Combined Aerobic and Isokinetic Strength Exercise Group
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Structured aerobic exercise (treadmill).
  Arms: Arm 2; Arm 4
Behavioral: Exercise — Structured isokinetic strength exercise (dynameter).
  Arms: Arm 3; Arm 4

SUMMARY:
This study will determine the type and combination of exercise needed to rehabilitate the neuro-compromised diabetic Veteran. Guided exercise protocols may prove to be practical therapeutic options for the prophylactic management of diabetic subjects with neuropathy.

DETAILED DESCRIPTION:
Purpose: A single-site, randomized, blinded, prospective clinical trial is proposed to determine the significance of a combined isokinetic strength and aerobic exercise training program on the rehabilitation of peripheral nerve function in Type 2 diabetic veterans and non-veterans with neuropathy. Background and Significance: Obesity is a major factor in the increasing rates of diabetes and its related complications. Diabetes affects greater than 7% of the population. Veterans are at even greater risk, with approximately 16% currently receiving treatment at Department of Veterans Affairs Medical Centers for diabetes. More than half of affected veterans experience debilitating complications of diabetes, including peripheral neuropathy (PN). Exercise training, in combination with pharmacologic intervention, is now recognized as a cornerstone of management for diabetes. Therapeutic interventions currently available for the treatment of PN in diabetic patients are limited, however, to pain management and stringent glycemic control. Exercise is reported to significantly decrease peripheral nerve microvascular complications common among chronic diabetics. Our preliminary findings demonstrate that exercise intervention improves peripheral nerve function in the diabetic veteran with PN. Intervention strategies, such as proposed in this application, offer a unique and novel therapeutic option for the rehabilitation of the neuro-compromised Type 2 diabetic veterans and non-veterans. Methods & Research Plan: One-hundred subjects will be recruited for this 24-week study. Subjects each will be randomly assigned to aerobic, isokinetic strength training, combined aerobic and strength training, or non-exercise (control) intervention groups. Isokinetic strength training (Biodex System 3), aerobic exercise training (treadmill), or the combination of strength and aerobic training will be administered 3x per week for the initial 12 weeks. Control subjects will receive 12 clinical visits over the course of the initial 12 weeks. The effects of exercise training type, compared with control subjects, on recovery of peripheral nerve function will be rigorously determined from baseline, 12- and 24-week testing using electrodiagnostic primary outcome measures, Quantitative Sensory Testing, and a battery of validated qualitative and quantitative secondary outcome measures that include an incremental symptom-limited treadmill test, peak torque, Total Neuropathy Score, visual analogue pain scale, and quality of life SF-36V Health Survey. Sustainability of effect will be determined at 24-weeks.The individual effects of exercise training type, compared with control subjects, on tissue oxygenation will be determined from baseline, 12- and 24-week testing by non-invasive quantitated infrared spectroscopy using an InSpectraTM Tissue Spectrometer. Expected Outcomes: This study will objectively and critically determine the type and combination of exercise needed to rehabilitate the neuro-compromised diabetic Veteran. Guided exercise protocols may prove to be practical therapeutic options for the prophylactic management of diabetic subjects with neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus
* stable blood glucose control
* clinical findings consistent with length-dependent sensorimotor polyneuropathy, stage N2a

Exclusion Criteria:

* foot ulceration
* unstable heart disease
* co-morbid conditions limiting exercise
* disorders of the central nervous system causing weakness or sensory loss
* received treatment with medications known to have neuropathy as a prominent side effect including vincristine, vinblastine, cis-platin, and paclitaxel
* medical conditions that may be associated with neuropathies such as alcoholism, liver disease, kidney disease, toxic exposure, vitamin deficiency, autoimmune disorders, cancer, or hypothyroidism

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01-14 (Actual); Primary Completion 2014-11-14 (Actual); Study Completion 2014-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Stubbs, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

REFERENCES:
- [Derived] Stubbs EB Jr, Fisher MA, Miller CM, Jelinek C, Butler J, McBurney C, Collins EG. Randomized Controlled Trial of Physical Exercise in Diabetic Veterans With Length-Dependent Distal Symmetric Polyneuropathy. Front Neurosci. 2019 Feb 11;13:51. doi: 10.3389/fnins.2019.00051. eCollection 2019. PMID 30804739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Edward Hines Jr. VA Hospital from January 2010-May 2014.
Pre-assignment Details: Prior to group randomization, all consenting subjects underwent two separate symptom-limited treadmill stress tests to unmask potentially life-threatening indolent cardiac and/or respiratory disease limitations
Groups:
- Sedentary: Sedentary Control Group
- Aerobic Exercise: Structured aerobic exercise (treadmill).
- Strength Exercise: Structured isokinetic strength exercise (dynameter).
- Combined Aerobic and Strength: Structured aerobic exercise (treadmill) plus structured isokinetic strength exercise (dynameter).
Period: Overall Study
Arm/Group | Sedentary | Aerobic Exercise | Strength Exercise | Combined Aerobic and Strength
Started | 12 | 11 | 11 | 11
Completed | 8 | 11 | 10 | 7
Not Completed | 4 | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Population studied are US Veterans and civilians diagnosed with long-standing (9-13y) type 2 diabetes mellitus with length-dependent distal polyneuropathy. Subjects were randomly assigned to either Sedentary, Aerobic Exercise, Strength Exercise, or a combination of Aerobic and Strength Exercise using "Research Randomizer" in blocks of 8.
Groups:
- Combined Aerobic and Strength: Structured aerobic exercise (treadmill).plus structured isokinetic strength exercise (dynameter).
- Total: Total of all reporting groups
Arm/Group | Sedentary | Aerobic Exercise | Strength Exercise | Combined Aerobic and Strength | Total
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (7.0) | 61.9 (8.3) | 64.2 (9.5) | 63.0 (6.6) | 62.5 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 2
  Male | 12 | 10 | 11 | 10 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 7 | 6 | 7 | 26
  African American | 6 | 3 | 4 | 3 | 16
  Hispanic | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: Count of Participants]
  United States | 12 | 11 | 11 | 11 | 45

OUTCOME MEASURES:

1. Primary Outcome: Sural Nerve Amplitude
Description: Maximal responses were obtained using percutaneous electrical stimuli. Sensory nerve action potentials were recorded from sural (antidromic), median (antidromic to second digit), and ulnar nerves (antidromic to fifth digit).To minimize inter-examiner variability and maximize neurophysiologic test/retest reliability, the same experienced neurologist conducted all nerve conduction studies on days separate from all other testing activities. A dedicated TECA Synergy electromyograph system was used for all nerve conduction studies. The patients dominant side was chosen. In patients with definable differences between the two sides, the side with the most prominent clinical findings was chosen. In all cases, the same limb was used for all three (baseline, 12-weeks, 24-weeks) conduction studies.
Time Frame: Baseline, 12, and 24 weeks
Population: Subjects withdrew from study prior to 3 month (# 3) and 6 month (# 1) evaluation. Subjects were withdrawn from study by principal/ co-principal investigator prior to 3 month (# 2) and 6 month (# 1) evaluation. Total difference = 7 at 6 month evaluation. Data shown include responders and non-responders.
Measure: Mean (Standard Deviation); unit: uV
Groups:
- Sedentary Control Group: Sedentary Control Group
- Aerobic Exercise Group: Aerobic Exercise Group
  Exercise: Structured aerobic exercise (treadmill).
- Strength Exercise Group: Strength Exercise Group
  Exercise: Structured isokinetic strength exercise (dynameter).
- Combined Aerobic and Strength Exercise Group: Combined Aerobic and Isokinetic Strength Exercise Group
  Exercise: Structured aerobic exercise (treadmill).
  Exercise: Structured isokinetic strength exercise (dynameter).
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
uV
  Baseline | 1.22 (2.93) | 2.37 (4.20) | 0.88 (2.92) | 0.86 (1.93)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 2.88 (3.84) | 1.49 (2.58) | 0.58 (1.83) | 1.21 (2.41)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 2.17 (3.28) | 2.93 (3.39) | 0.86 (2.72) | 0.65 (1.84)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.49, ANOVA — Tukey's multiple comparisons test; Comparison to baseline values
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.82, ANOVA — Tukey's multiple comparisons test
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.96, ANOVA — Tukey's multiple comparisons test
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.93, ANOVA — Tukey's multiple comparisons test
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.63, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wk; Test type: Superiority; p = 0.31, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wk; Test type: Superiority; p = 0.28, ANOVA

2. Primary Outcome: Sural Nerve Latency
Description: as for outcome 1
Time Frame: Baseline, 12 wks, 24 wks
Population: Subjects withdrew from study prior to 3 month (# 3) and 6 month (# 1) evaluation Subjects were withdrawn from study by principal/ co-principal investigator prior to 3 month (# 2) and 6 month (# 1) evaluation. Total difference = 7 at 6 month evaluation. Data shown include responders and non-responders.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
ms
  Baseline | 0.61 (1.43) | 1.01 (1.73) | 0.39 (1.3) | 0.64 (1.43)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 1.41 (1.83) | 1.04 (1.79) | 0.42 (1.33) | 0.89 (1.76)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 1.26 (1.91) | 1.57 (1.86) | 0.4 (1.26) | 0.48 (1.34)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.53, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.93, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.80, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.63, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wk; Test type: Superiority; p = 0.31, ANOVA

3. Primary Outcome: Sural Nerve Conduction Velocity
Description: as for outcome 1
Time Frame: Baseline, 12 wks, 24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Strength Exercise Group: Isokinetic Strength Exercise Group
  Exercise: Structured isokinetic strength exercise (dynameter).
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
m/s
  baseline | 6.21 (14.5) | 11.1 (19.26) | 3.27 (10.85) | 7.35 (16.38)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 16.46 (21.32) | 10.55 (18.24) | 3.73 (11.8) | 8.62 (17.14)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 12.38 (18.63) | 18.54 (21.48) | 3.88 (12.27) | 5.34 (15.10)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.39, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.98, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.70, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.45, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.22, ANOVA

4. Primary Outcome: Tibial Nerve Amplitude
Description: Maximal responses were obtained using percutaneous electrical stimuli. Distal motor nerve evoked compound muscle action potential (CMAP) potentials were recorded from tibial and peroneal nerves.To minimize inter-examiner variability and maximize neurophysiologic test/retest reliability, the same experienced neurologist conducted all nerve conduction studies on days separate from all other testing activities. A dedicated TECA Synergy electromyograph system was used for all nerve conduction studies. The patients dominant side was chosen. In patients with definable differences between the two sides, the side with the most prominent clinical findings was chosen. In all cases, the same limb was used for all three (baseline, 12-weeks, 24-weeks) conduction studies.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
mV
  Baseline | 2.97 (3.13) | 3.71 (3.91) | 3.35 (3.43) | 4.71 (3.73)
  12 wks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 wks | 3.26 (3.32) | 3.03 (3.39) | 3.73 (3.93) | 3.59 (3.75)
  24 wks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 wks | 3.48 (3.62) | 3.46 (3.57) | 3.90 (4.04) | 3.33 (3.68)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.98, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.90, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.97, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.78, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.63, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wk; Test type: Superiority; p = 0.97, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.99, ANOVA

5. Primary Outcome: Tibial Nerve Latency
Description: as for outcome 4
Time Frame: Baseline, 12 weeks, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
ms
  Baseline | 4.37 (1.5) | 5.03 (0.72) | 4.43 (1.56) | 4.11 (1.47)
  12 wks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 wks | 4.15 (1.62) | 4.65 (1.62) | 4.28 (1.65) | 4.29 (1.78)
  24 wks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 wks | 4.41 (1.7) | 5.25 (0.57) | 4.40 (2.43) | 5.29 (1.76)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.94, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.69, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.98, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.97, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.45, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.91, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.51, ANOVA

6. Primary Outcome: Tibial Nerve Conduction Velocity
Description: as for outcome 4
Time Frame: Baseline, 12 weeks, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
m/s
  Baseline | 31.81 (10.42) | 33.15 (4.01) | 30.0 (10.29) | 30.43 (10.58)
  12 wks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 wks | 32.56 (12.51) | 30.77 (11.05) | 30.64 (11.52) | 31.08 (11.9)
  24 wks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 wks | 30.22 (13.43) | 34.22 (4.17) | 28.51 (15.85) | 31.73 (5.58)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.72, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.85, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.98, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.68, ANOVA

7. Primary Outcome: Sensory Median Nerve Amplitude
Description: as for outcome 1
Time Frame: Baseline, 12, and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
uV
  Baseline | 3.14 (4.44) | 5.55 (8.12) | 6.91 (4.61) | 7.18 (6.88)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 2.41 (3.23) | 6.00 (9.71) | 6.26 (4.17) | 6.10 (6.99)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 4.52 (4.47) | 6.06 (8.12) | 4.97 (4.41) | 4.31 (6.56)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.91, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.94, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.93, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.38, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.51, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.94, ANOVA

8. Primary Outcome: Sensory Median Nerve Latency
Description: as for outcome 1
Time Frame: Baseline, 12wks, 24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Aerobic Exercise Group: Structured aerobic exercise (treadmill).
- Strength Exercise Group: Structured isokinetic strength exercise (dynameter).
- Combined Aerobic and Strength Exercise Group: Structured aerobic exercise (treadmill) plus structured isokinetic strength exercise (dynameter).
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
ms
  Baseline | 1.66 (2.05) | 1.76 (2.06) | 3.36 (1.75) | 2.26 (1.83)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 1.54 (1.99) | 2.00 (2.36) | 3.15 (1.75) | 2.19 (2.11)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 2.72 (2.07) | 2.44 (2.43) | 2.87 (2.03) | 1.81 (1.99)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.97, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.96, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.16, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.37, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.75, ANOVA

9. Primary Outcome: Sensory Median Nerve Conduction Velocity
Description: as for outcome 1
Time Frame: Baseline, 12 wks, 24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
m/s
  Baseline | 18.95 (23.83) | 20.34 (23.59) | 35.05 (18.19) | 30.49 (25.08)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 18.18 (23.73) | 19.04 (22.17) | 35.73 (19.8) | 23.64 (22.93)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 30.00 (22.74) | 22.90 (22.63) | 29.76 (21.03) | 22.88 (25.21)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.81, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.28, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.28, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.83, ANOVA

10. Primary Outcome: Sensory Ulnar Nerve Amplitude
Description: as for outcome 1
Time Frame: Baseline, 12 wks, 24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
uV
  Baseline | 4.48 (4.08) | 4.95 (5.10) | 5.60 (7.63) | 7.75 (5.77)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 4.68 (4.84) | 4.44 (6.71) | 3.87 (5.41) | 8.49 (5.89)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 6.08 (5.12) | 4.12 (2.88) | 6.97 (6.17) | 8.68 (6.89)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.97, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.82, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.96, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.55, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.31, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.32, ANOVA

11. Primary Outcome: Sensory Ulnar Nerve Latency
Description: as for outcome 1
Time Frame: Baseline, 12 wks, 24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
ms
  Baseline | 2.25 (1.73) | 1.78 (1.72) | 1.50 (1.76) | 2.46 (1.26)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 1.82 (1.58) | 1.49 (1.75) | 1.24 (1.64) | 2.36 (1.39)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 2.56 (1.47) | 2.53 (1.66) | 2.36 (1.66) | 2.24 (1.45)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.81, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.92, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.93, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.50, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.47, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.97, ANOVA

12. Primary Outcome: Sensory Ulnar Nerve Conduction Velocity
Description: as for outcome 1
Time Frame: Baseline, 12 wks, 24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
m/s
  Baseline | 29.29 (22.19) | 24.68 (23.94) | 20.61 (24.06) | 39.27 (20.14)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 23.64 (25.03) | 20.59 (23.99) | 19.81 (25.83) | 36.40 (20.87)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 34.10 (19.48) | 30.91 (20.12) | 31.54 (22.09) | 36.06 (23.31)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.83, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.91, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.95, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.26, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.42, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.95, ANOVA

13. Primary Outcome: Peroneal Nerve Amplitude
Description: as for outcome 4
Time Frame: Baseline, 12 wks, 24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
mV
  Baseline | 2.16 (2.17) | 2.33 (2.01) | 1.89 (1.68) | 2.79 (1.91)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 1.89 (2.27) | 1.55 (1.51) | 1.43 (1.35) | 2.52 (1.47)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 2.45 (2.72) | 1.70 (1.51) | 1.75 (1.73) | 2.71 (1.97)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.96, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.53, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.79, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.94, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.75, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.51, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.63, ANOVA

14. Primary Outcome: Peroneal Nerve Latency
Description: as for outcome 4
Time Frame: Baseline, 12 wks, 24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
ms
  Baseline | 4.69 (2.58) | 4.93 (1.95) | 4.96 (1.88) | 4.65 (1.88)
  12 weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12 weeks | 4.49 (2.72) | 4.85 (1.72) | 4.52 (2.46) | 5.06 (2.17)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 4.69 (3.10) | 4.63 (1.65) | 5.28 (2.14) | 4.68 (2.20)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluated within group across time; Test type: Superiority; p = 0.98, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluated within group across time; Test type: Superiority; p = 0.89, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.90, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.98, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.94, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.91, ANOVA

15. Primary Outcome: Peroneal Nerve Conduction Velocity
Description: as for outcome 4
Time Frame: Baseline, 12 wks, 24 wks
Population: Subjects withdrew from study prior to 3 month (# 3) and 6 month (# 1) evaluation Subjects were withdrawn from study by principal/ co-principal investigator prior to 3 month (# 2) and 6 month (# 1) evaluation. No data recorded for 1 Sedentary subject at 3 month evaluation. Data shown include responders and non-responders.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
m/s
  Baseline | 30.58 (14.92) | 32.01 (11.82) | 32.97 (13.59) | 33.33 (11.82)
  12 weeks: number analyzed (Participants) | 9 | 11 | 10 | 9
  12 weeks | 29.07 (16.98) | 32.56 (11.15) | 29.46 (16.19) | 33.86 (13.28)
  24 weeks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24 weeks | 29.41 (17.28) | 33.40 (11.56) | 31.06 (12.27) | 33.08 (13.69)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 0.98, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.84, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.96, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.86, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.92, ANOVA

16. Secondary Outcome: Symptom-Limited TMT Blood Glucose Response
Description: Changes in blood glucose in response to modified Bruce Protocol treadmill test (TMT)
Time Frame: Initial entry into study, 12 and 24 weeks
Population: Subj. withdrew from study prior to 3 mo. (#3) and 6 mo. (#1) eval. Subj. withdrawn from study by PI/co-PI prior to 3 month (#2) and 6 month (#1) eval. Total difference = 8 at 6 mo. eval. 1(Sed) had EMG @ 12 and 24 wks didn't receive clearance for TMT but to continue in other study activities. 1 (Sed) post 24 week EMG and withdrawn s/p hosp.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
mg/dl
  Baseline-Pre Exercise | 157.3 (49.5) | 188.6 (65.6) | 181.5 (48.9) | 180.7 (43.2)
  Baseline-Post Exercise | 129.3 (41.7) | 169.4 (46.0) | 138.5 (48.7) | 149.5 (46.1)
  12-weeks-Pre Exercise: number analyzed (Participants) | 9 | 11 | 9 | 8
  12-weeks-Pre Exercise | 188.7 (68.6) | 171.7 (47.9) | 170.6 (43.9) | 160.0 (51.2)
  12-weeks-Post Exercise: number analyzed (Participants) | 9 | 11 | 9 | 8
  12-weeks-Post Exercise | 127.3 (36.0) | 151.1 (41.4) | 147.2 (59.7) | 128.0 (28.7)
  24-weeks-Pre Exercise: number analyzed (Participants) | 7 | 11 | 9 | 7
  24-weeks-Pre Exercise | 163.9 (46.0) | 181.8 (62.9) | 187.9 (53.6) | 169.0 (48.9)
  24-weeks-Post Exercise: number analyzed (Participants) | 7 | 11 | 9 | 7
  24-weeks-Post Exercise | 143.6 (33.8) | 166.3 (57.9) | 161.9 (43.5) | 139.4 (45.9)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group pre- and post-test responses across time; Test type: Superiority; p = 0.03, t-test, 2 sided — Unpaired two-tailed t-test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group pre- and post-test responses across time; Test type: Superiority; p = 0.29, t-test, 2 sided — Unpaired two-tailed t-test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group pre- and post-test responses across time; Test type: Superiority; p = 0.36, t-test, 2 sided — Unpaired two-tailed t-test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group pre- and post-test responses across time; Test type: Superiority; p = 0.15, t-test, 2 sided — Unpaired two-tailed t-test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison of pre- and post-responses across groups at baseline; Test type: Superiority; p = 0.20, ANOVA — ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison of pre- and post-test responses across groups at 12 wks; Test type: Superiority; p = 0.51, ANOVA — ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison of pre- and post-test responses across groups at 24 wks; Test type: Superiority; p = 0.59, ANOVA — ANOVA

17. Secondary Outcome: Short Form-36V: Physical Component Score
Description: The short form-36Veterans (SF-36V) health survey questionnaire was used to measure health-related quality of life. This survey is comprised of eight subscales and two overall component scores, all of which have demonstrated high levels of internal consistency and discriminate validity when administered to groups of medically stable individuals. Patient aggregate responses for the eight distinct summary subscales and two component scores were compiled as a percentage of total points possible using the RAND 36-item health survey table. Data shown are expressed as a percentage of total possible score ranging from 0%-100% with 100% considered relatively good health and 0% considered poor health. Physical Component scores reflect perceived changes in physical health relative to the previous year.
Time Frame: Initial entry into study, 12 and 24 weeks
Population: Subj. withdrew from study prior to 3 mo. (#3) and 6 mo. (#1) eval. Subj. withdrawn from study by PI/coPI prior to 3 month (#2) and 6 month (#1) eval. Total difference = 8 at 6 mo. eval. 1(Sed) had EMG @ 12 and 24 wks didn't receive clearance for TMT but to continue in other study activities. 1 (Sed) post 24 week EMG and withdrawn s/p hosp.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedentary | Aerobic Exercise | Strength Exercise | Combined Aerobic and Strength
Number analyzed (Participants) | 12 | 11 | 11 | 11
score on a scale
  Baseline | 60.4 (29.1) | 52.3 (26.1) | 56.8 (25.2) | 59.1 (28.0)
  12-weeks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12-weeks | 57.5 (23.7) | 86.4 (17.2) | 65.0 (26.9) | 72.2 (29.2)
  24-weeks: number analyzed (Participants) | 9 | 11 | 10 | 7
  24-weeks | 58.3 (21.7) | 86.4 (17.2) | 77.5 (32.2) | 75.0 (32.3)
Statistical Analysis 1: Comparison: Sedentary; Evaluate within group across time; Test type: Superiority; p = 1.00, Kruskal-Wallis — Dunn's multiple comparisons
Statistical Analysis 2: Comparison: Aerobic Exercise; Evaluate within group across time; Test type: Superiority; p = 0.01, Kruskal-Wallis — Dunn's multiple comparisons
Statistical Analysis 3: Comparison: Strength Exercise; Evaluate within group across time; Test type: Superiority; p = 1.00, Kruskal-Wallis — Dunn's multiple comparisons
Statistical Analysis 4: Comparison: Combined Aerobic and Strength; Evaluate within group across time; Test type: Superiority; p = 0.98, Kruskal-Wallis — Dunn's multiple comparisons
Statistical Analysis 5: Comparison: Sedentary vs Aerobic Exercise vs Strength Exercise vs Combined Aerobic and Strength; Comparison across groups at baseline; Test type: Superiority; p = 0.96, Kruskal-Wallis
Statistical Analysis 6: Comparison: Sedentary vs Aerobic Exercise vs Strength Exercise vs Combined Aerobic and Strength; Comparison across groups at 12-wks; Test type: Superiority; p = 0.06, Kruskal-Wallis
Statistical Analysis 7: Comparison: Sedentary vs Aerobic Exercise vs Strength Exercise vs Combined Aerobic and Strength; Comparison across groups at 24-wks; Test type: Superiority; p = 0.14, Kruskal-Wallis

18. Secondary Outcome: Voluntary Duration of Symptom-Limited TMT
Description: Total time subjects voluntarily exercised while undergoing a modified Bruce Protocol treadmill test (TMT)
Time Frame: baseline, 12-wks, 24-wks
Population: Subj. withdrew from study prior to 3 mo. (#3) and 6 mo. (#2) eval. Subj. withdrawn from study by PI/coPI prior to 3 month (#2) and 6 month (#1) eval. Total difference = 8 at 6 mo. eval. 1(Sed) had EMG @ 12 and 24 wks didn't receive clearance for TMT but to continue in other study activities. 1 (Sed) fell post 24 week EMG and withdrawn s/p hosp.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
minutes
  Baseline | 10.8 (3.5) | 11.9 (2.2) | 8.8 (2.9) | 11.0 (3.5)
  12-weeks: number analyzed (Participants) | 9 | 11 | 9 | 9
  12-weeks | 10.7 (3.8) | 13.4 (2.5) | 9.3 (3.0) | 13.0 (4.4)
  24-weeks: number analyzed (Participants) | 7 | 11 | 9 | 6
  24-weeks | 11.4 (3.9) | 13.3 (2.9) | 9.0 (2.9) | 14.2 (2.8)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.36, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.93, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.46, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.14, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12 wks; Test type: Superiority; p = 0.05, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24 wks; Test type: Superiority; p = 0.01, ANOVA

19. Secondary Outcome: Symptom-Limited TMT Maximum Heart Rate
Description: Peak heart rate achieved while undergoing a modified Bruce Protocol treadmill test (TMT)
Time Frame: baseline, 12-wks, 24-wks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: beats per min
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
beats per min
  Baseline | 128.5 (31.9) | 141.5 (18.9) | 135.5 (26.6) | 146.0 (23.3)
  12-weeks: number analyzed (Participants) | 9 | 11 | 9 | 9
  12-weeks | 125.8 (37.9) | 143.1 (21.6) | 126.0 (24.9) | 135.9 (25.4)
  24-weeks: number analyzed (Participants) | 7 | 11 | 9 | 6
  24-weeks | 127.4 (29.3) | 140.5 (24.1) | 129.3 (21.4) | 143.3 (16.8)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 0.98, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.98, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.67, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.55, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.40, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12 wks; Test type: Superiority; p = 0.47, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24 wks; Test type: Superiority; p = 0.43, ANOVA

20. Secondary Outcome: Symptom-Limited TMT Maximum Systolic Blood Pressure
Description: Peak systolic BP achieved while undergoing a modified Bruce Protocol treadmill test (TMT)
Time Frame: Baseline, 12-wk, 24-wk
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
mmHg
  Baseline | 190.5 (26.5) | 189.3 (26.7) | 196.3 (25.5) | 188.4 (20.4)
  12-weeks: number analyzed (Participants) | 9 | 11 | 9 | 9
  12-weeks | 196.0 (19.8) | 185.8 (17.8) | 200.0 (28.6) | 184.0 (29.8)
  24-weeks: number analyzed (Participants) | 7 | 11 | 9 | 6
  24-weeks | 179.1 (13.9) | 180.7 (20.6) | 193.1 (21.4) | 185.3 (9.9)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 0.84, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.93, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.94, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.94, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.88, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12 wks; Test type: Superiority; p = 0.48, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24 wks; Test type: Superiority; p = 0.38, ANOVA

21. Secondary Outcome: Symptom-Limited TMT Maximum Minute Ventilation (VE)
Description: Peak volume of air exchanged per minute achieved while undergoing a modified Bruce Protocol treadmill test (TMT)
Time Frame: Baseline, 12-wks, 24-wks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liters/min
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
liters/min
  Baseline | 62.9 (15.3) | 63.5 (18.8) | 54.3 (12.9) | 62.0 (13.3)
  12-weeks: number analyzed (Participants) | 9 | 11 | 9 | 9
  12-weeks | 59.9 (10.6) | 67.0 (22.2) | 60.6 (12.1) | 62.4 (15.5)
  24-weeks: number analyzed (Participants) | 7 | 11 | 9 | 6
  24-weeks | 57.4 (13.1) | 73.2 (27.3) | 56.4 (12.4) | 68.8 (13.1)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 0.87, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.93, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.51, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.89, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.46, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12 wks; Test type: Superiority; p = 0.72, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24wks; Test type: Superiority; p = 0.22, ANOVA

22. Secondary Outcome: Symptom-Limited TMT Maximum Oxygen Uptake (VO2)
Description: Peak Oxygen uptake achieved while undergoing a modified Bruce Protocol treadmill test (TMT)
Time Frame: Baseline, 12-wks, 24-wks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
ml/min/kg
  Baseline | 17.4 (3.9) | 18.9 (4.2) | 16.5 (3.8) | 18.9 (3.6)
  12-weeks: number analyzed (Participants) | 9 | 11 | 9 | 9
  12-weeks | 17.0 (4.6) | 18.7 (5.1) | 17.2 (3.0) | 18.9 (4.7)
  24-weeks: number analyzed (Participants) | 7 | 11 | 9 | 6
  24-weeks | 18.2 (4.6) | 19.3 (5.3) | 16.5 (2.2) | 21.8 (3.4)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 0.98, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.99, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.87, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.95, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.39, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.59, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.29, ANOVA

23. Secondary Outcome: Maximum Respiratory Exchange Ratio (RER) During TMT
Description: Peak RER achieved while undergoing a modified Bruce Protocol treadmill test (TMT). This is a mathematical ratio of maximally achieved (peak) VCO2 divided by maximally achieved (peak) VO2.
Time Frame: Baseline, 12-wks, 24-wks
Population: Subj. withdrew from study prior to 3 mo. (#3) and 6 mo. (#2) eval. Subj. withdrawn from study by PI/coPI prior to 3 month (#2) and 6 month (#1) eval. Total difference = 8 at 6 mo. eval. 1(Sed) had EMG @ 12 and 24 wks didn't receive clearance for TMT but to continue in other study activities. 1 (Sed) post 24 week EMG and withdrawn s/p hosp.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
ratio
  Baseline | 1.2 (0.1) | 1.2 (0.2) | 1.1 (0.1) | 1.1 (0.1)
  12-weeks: number analyzed (Participants) | 9 | 11 | 9 | 9
  12-weeks | 1.2 (0.1) | 1.2 (0.1) | 1.2 (0.1) | 1.2 (0.1)
  24-weeks: number analyzed (Participants) | 7 | 11 | 9 | 6
  24-weeks | 1.2 (0.1) | 1.2 (0.1) | 1.1 (0.1) | 1.1 (0.0)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 0.97, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.09, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.05, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.11, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.41, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.03, ANOVA

24. Secondary Outcome: Symptom-Limited TMT Maximum Carbon Dioxide Expelled (VCO2)
Description: Peak Carbon Dioxide expelled achieved while undergoing a modified Bruce Protocol treadmill test (TMT)
Time Frame: Baseline, 12-wks, 24-wks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
ml/min/kg
  Baseline | 20.4 (4.7) | 22.0 (6.4) | 18.9 (5.4) | 20.7 (4.1)
  12-weeks: number analyzed (Participants) | 9 | 11 | 9 | 8
  12-weeks | 19.7 (4.9) | 21.9 (7.3) | 19.9 (3.9) | 23.7 (7.4)
  24-weeks: number analyzed (Participants) | 7 | 11 | 9 | 7
  24-weeks | 20.2 (6.3) | 22.5 (7.1) | 18.7 (3.4) | 23.4 (4.8)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 0.95, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.87, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.48, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.58, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.50, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.33, ANOVA

25. Secondary Outcome: Symptom-Limited TMT Maximum METS Achieved (MET)
Description: Peak metabolic rate equivalents (METS) achieved while undergoing a modified Bruce Protocol treadmill test (TMT). One MET is defined as the metabolic rate observed at rest, quantified as resting oxygen consumption of 250 ml/min (Male) or 200 ml /min (female). A value of 5 METS would represent a metabolic rate that is 5x that at rest and is considered an indicator of how hard a given individual is exercising. Data shown are expressed as a ratio at peak of exercise of oxygen consumed relative to normalized values for men or women at rest.
Time Frame: Baseline, 12-wks, 24-wks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
ratio
  Baseline | 5.0 (1.1) | 5.4 (1.2) | 4.7 (1.1) | 5.4 (1.0)
  12-weeks: number analyzed (Participants) | 9 | 11 | 9 | 8
  12-weeks | 4.9 (1.3) | 5.4 (1.4) | 4.9 (0.9) | 5.6 (1.3)
  24-weeks: number analyzed (Participants) | 7 | 11 | 9 | 7
  24-weeks | 5.2 (1.3) | 5.5 (1.5) | 4.8 (0.6) | 5.9 (1.2)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 0.98, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.88, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.93, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.38, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.55, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.37, ANOVA

26. Secondary Outcome: Short Form-36V: Mental Component Score
Description: The short form-36Veterans (SF-36V) health survey questionnaire was used to measure health-related quality of life. This survey is comprised of eight subscales and two overall component scores, all of which have demonstrated high levels of internal consistency and discriminate validity when administered to groups of medically stable individuals. Patient aggregate responses for the eight distinct summary subscales and two component scores were compiled as a percentage of total points possible using the RAND 36-item health survey table. Data shown are expressed as a percentage of total possible score ranging from 0%-100% with 100% considered relatively good health and 0% considered poor health. Mental Component scores reflect perceived changes in emotional health relative to the previous year.
Time Frame: initial entry into study, and at 12-wks and 24-wks
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Combined Aerobic and Strength Exercise Group: Structured aerobic exercise (treadmill).plus structured isokinetic strength exercise (dynameter).
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
score on a scale
  Baseline | 68.8 (32.2) | 63.6 (30.3) | 59.1 (25.7) | 61.4 (28.2)
  12-wks: number analyzed (Participants) | 10 | 11 | 10 | 9
  12-wks | 65.0 (17.5) | 72.7 (20.8) | 60.0 (26.9) | 72.2 (26.4)
  24-wks: number analyzed (Participants) | 9 | 11 | 10 | 7
  24-wks | 75.0 (21.7) | 75.0 (19.4) | 67.5 (33.4) | 75.0 (25.0)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 1.00, Kruskal-Wallis — Dunn's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, Kruskal-Wallis — Dunn's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, Kruskal-Wallis — Dunn's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, Kruskal-Wallis — Dunn's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.81, Kruskal-Wallis
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12-wks; Test type: Superiority; p = 0.60, Kruskal-Wallis
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24-wks; Test type: Superiority; p = 0.99, Kruskal-Wallis

27. Other Pre Specified Outcome: Height
Description: Height of subjects upon entry into study
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
cm | 178.1 (5.8) | 181.0 (8.6) | 179.9 (5.3) | 177.4 (7.1)
Statistical Analysis 1: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.59, ANOVA

28. Other Pre Specified Outcome: Weight
Description: Weight of subjects at baseline, 12-weeks, and 24-weeks
Time Frame: Baseline, 12-wks, 24-wks
Population: Subjects withdrew from study prior to 3 month (# 3) and 6 month (# 2) evaluation Subjects were withdrawn from study by principal/ co-principal investigator prior to 3 month (# 2) and 6 month (# 1) evaluation. Total difference = 8 at 6 month evaluation.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
kg
  Baseline | 104.7 (14.4) | 109.9 (19.7) | 102.6 (16.3) | 101.3 (14.4)
  12-wks: number analyzed (Participants) | 11 | 11 | 11 | 9
  12-wks | 103.7 (12.9) | 109.8 (18.5) | 102.9 (17) | 97.1 (9.7)
  24-wks: number analyzed (Participants) | 9 | 11 | 10 | 8
  24-wks | 100.5 (10.5) | 109.8 (18.3) | 103.8 (17.6) | 98.4 (10.7)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 0.98, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.72, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.62, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12 wks; Test type: Superiority; p = 0.33, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24 wks; Test type: Superiority; p = 0.38, ANOVA

29. Other Pre Specified Outcome: Body Mass Index (BMI)
Description: BMI is calculated as a ratio of subject body mass (kg) divided by the square of subject height (m).
Time Frame: Baseline, 12-wk, 24-wk
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
kg/m^2
  Baseline | 32.9 (3.5) | 33.4 (5.4) | 31.5 (4.1) | 32.4 (6.3)
  12-wk: number analyzed (Participants) | 11 | 11 | 11 | 9
  12-wk | 32.3 (2.8) | 33.4 (5.0) | 31.6 (4.2) | 30.8 (4.0)
  24-wk: number analyzed (Participants) | 9 | 11 | 9 | 8
  24-wk | 31.5 (2.6) | 33.4 (4.9) | 31.9 (4.3) | 31.5 (3.8)
Statistical Analysis 1: Comparison: Sedentary Control Group; Evaluate within group across time; Test type: Superiority; p = 0.88, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 3: Comparison: Aerobic Exercise Group vs Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 1.00, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 4: Comparison: Combined Aerobic and Strength Exercise Group; Evaluate within group across time; Test type: Superiority; p = 0.76, ANOVA — Tukey's multiple comparisons test:
Statistical Analysis 5: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.82, ANOVA
Statistical Analysis 6: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 12 wks; Test type: Superiority; p = 0.53, ANOVA
Statistical Analysis 7: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at 24 wks; Test type: Superiority; p = 0.68, ANOVA

30. Other Pre Specified Outcome: Duration of Diabetes Mellitus
Description: Duration, in years, since first diagnosed with Diabetes Mellitus upon entry into study
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
years | 12.6 (11.1) | 10.9 (4.1) | 10.1 (6.7) | 8.9 (6.3)
Statistical Analysis 1: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.70, ANOVA

31. Other Pre Specified Outcome: HbA1C Laboratory Values
Description: Laboratory values of subject HbA1C levels at Baseline, 12-wk, 24-wk
Time Frame: Baseline, 12-wk, 24-wk
Population: A1c testing was performed prior to EMG evaluation so there are 2/4 additional values for 3/6 month numbers of subjects than is reflected in the statement regarding subject withdrawal in the EMG sections. Total difference = 6 at 6 month evaluation.
Measure: Mean (Standard Deviation); unit: percentage of Hb
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
percentage of Hb
  Baseline | 7.8 (0.5) | 8.0 (1.0) | 8.0 (1.0) | 7.2 (0.7)
  12-wk: number analyzed (Participants) | 12 | 11 | 11 | 9
  12-wk | 7.7 (1.0) | 8.0 (1.5) | 7.4 (1.0) | 7.3 (1.0)
  24-wk: number analyzed (Participants) | 9 | 11 | 10 | 9
  24-wk | 7.2 (1.1) | 7.9 (1.3) | 8.0 (1.2) | 7.1 (0.7)

32. Other Pre Specified Outcome: Triglyceride Laboratory Values
Description: Laboratory triglyceride values at baseline entry into study
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
mg/dL | 157.7 (84.5) | 125.0 (57.1) | 144.5 (68.2) | 162.0 (60)
Statistical Analysis 1: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.59, ANOVA

33. Other Pre Specified Outcome: Cholesterol Laboratory Values
Description: Laboratory total cholesterol, HDL-cholesterol, and LDL-cholesterol levels at baseline entry into study
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
mg/dL
  Total Cholesterol | 139.3 (25.1) | 156.4 (36.2) | 158.5 (39.7) | 159.9 (48.7)
  HDL-Cholesterol | 41.4 (29.0) | 42.8 (13.5) | 40.7 (14.0) | 38.4 (4.8)
  LDL-Cholesterol | 68.4 (23.3) | 88.6 (31.2) | 89.0 (42.5) | 89.2 (48.0)
Statistical Analysis 1: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.45, ANOVA

34. Other Pre Specified Outcome: Creatinine Laboratory Values
Description: Laboratory creatinine values at baseline entry into study
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
mg/dL | 1.1 (0.2) | 1.0 (0.1) | 0.9 (0.1) | 1.0 (0.2)
Statistical Analysis 1: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.04, ANOVA

35. Other Pre Specified Outcome: Blood Urea Nitrogen (BUN) Laboratory Values
Description: Laboratory Blood Urea Nitrogen levels at baseline entry into study
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
mg/dL | 17.0 (5.5) | 19.0 (5.9) | 16.5 (6.7) | 17.8 (5.6)
Statistical Analysis 1: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.77, ANOVA

36. Other Pre Specified Outcome: Aspartate Aminotransferase Laboratory Values
Description: Laboratory values for Aspartate Aminotransferase (AST) at baseline entry into study
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units/L
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
units/L | 20.8 (5.6) | 13.5 (6.3) | 19.5 (9.6) | 23.6 (15.2)
Statistical Analysis 1: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.12, ANOVA

37. Other Pre Specified Outcome: Thyroid Stimulating Hormone Laboratory Values
Description: Laboratory values for Thyroid Stimulating Hormone (TSH) at baseline entry into study
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
uIU/mL | 1.3 (0.6) | 1.8 (0.9) | 2.0 (1.6) | 1.8 (0.7)
Statistical Analysis 1: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.42, ANOVA

38. Other Pre Specified Outcome: Age
Description: Age of participants at entry into study.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Sedentary Control Group | Aerobic Exercise Group | Strength Exercise Group | Combined Aerobic and Strength Exercise Group
Number analyzed (Participants) | 12 | 11 | 11 | 11
years | 61.0 (7.0) | 61.9 (8.3) | 64.2 (9.5) | 63.0 (6.6)
Statistical Analysis 1: Comparison: Sedentary Control Group vs Aerobic Exercise Group vs Strength Exercise Group vs Combined Aerobic and Strength Exercise Group; Comparison across groups at baseline; Test type: Superiority; p = 0.79, ANOVA

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Combined Aerobic and Strength: Structured aerobic exercise (treadmill) and structured isokinetic strength exercise (dynameter).
Arm/Group | Sedentary | Aerobic Exercise | Strength Exercise | Combined Aerobic and Strength
All-Cause Mortality (participants affected / at risk) | 6/12 | 4/11 | 4/11 | 5/11
Serious Adverse Events (participants affected / at risk) | 6/12 | 4/11 | 4/11 | 5/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedentary (N=12) | Aerobic Exercise (N=11) | Strength Exercise (N=11) | Combined Aerobic and Strength (N=11)
4 years 6 months (Surgical and medical procedures) | 6 (11) | 4 (4) | 4 (9) | 5 (9)

LIMITATIONS AND CAVEATS:
Chronic type 2 diabetic patient population with advanced complications, including peripheral neuropathy, presented with unanticipated highly variable baseline measures that markedly diminished the studies statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2009-10-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT00955201/Prot_SAP_ICF_000.pdf